CLINICAL TRIAL: NCT01473277
Title: Intra-articular Injection of Botulinum Toxin Type A in Hemiplegic Shoulder Pain: a Multicentric, Double Blind Randomised, Versus Steroid Study
Brief Title: Botulinum Toxin Type A (BT-A) in Hemiplegic Shoulder Pain Versus Steroid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Foundation Institute San Raffaele G. Giglio of Cefalù (Other)
Collaborators: Ospedale di Brunico (Unknown); Fondazione Salvatore Maugeri (Other); IRCCS San Camillo, Venezia, Italy (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Giuseppe Galardi, Direttore Unità Operativa di Riabilitazione, The Foundation Institute San Raffaele G. Giglio of Cefalù
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-004682-32
Record Dates: First submitted 2011-11-07; First posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Stroke; Hemiparesis; Shoulder Pain
Keywords: Hemiplegic shoulder pain; Botulinum toxin type A (BT-A); Steroid; Intra-articular injection; Pain score of 45 or greater on a 0-100 mm VAS; Duration of HSP for at least one month; Pain refractoriness to conventional treatment
MeSH Terms: conditions — Stroke; Paresis; Shoulder Pain | interventions — abobotulinumtoxinA; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BT-A (Dysport 500U) (Active Comparator)
  Interventions: Drug: BT-A (Dysport 500U), Triamcinolone acetonide
- Triamcinolone acetonide (Active Comparator)
  Interventions: Drug: BT-A (Dysport 500U), Triamcinolone acetonide

INTERVENTIONS:
Drug: BT-A (Dysport 500U), Triamcinolone acetonide — All patients will be randomize to receive an intra-articular injection of BT-A (Dysport 500U) or triamcinolone acetonide (40 mg). Both drugs will be reconstituted with 2.0 ml of saline. Both drugs will be injected in the glenohumeral joint with a standard posterior approach. The time of the intra-articular injection od BT-A or steroid will be considered the "time zero" for each patient. The primary and secondary efficacy variables will be evaluated in all patients at 1 week, 2 weeks, 4 weeks, 3 months and 6 months after the treatment.

SUMMARY:
The aim of this study is to confirm the efficacy and safety of the intra-articular injection of BT-A in a multicentric double blind randomised study. For this purpose intra-articular injection of BT-A will be compared with the intra-articular steroid injection that is the current "gold standard" for the treatment of HSP.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common complications of stroke. In fact, it occurs up to 70% of stroke victims. Post-stroke shoulder pain impacts negatively on daily activities. Moreover, it interferes with the rehabilitation process, is related to poor quality of life and has been associated to a worse outcome and to prolonged hospitalization.The aetiology of post-stroke HSP is uncertain, although it has been associated with various factors: joint disorders, capsulitis adhesive, subluxation of the head of the humerus, rotator cuff tendons injuries and spasticity of surrounding muscles. Clinicians use a wide variety of approaches to treat post-stroke HSP, although none has yet been proven effective. Correct positioning and careful handling of the hemiplegic limb are believed to prevent HSP. Physiotherapy alone does not seem to be effective for this complication. Capsulitis adhesive can be successfully treated with corticosteroid injections in the shoulder. However, despite many randomized controlled trials of corticosteroid injections for shoulder pain, their effects remain controversial. The large number of interventions and the lack of consensus about their effectiveness suggest that the aetiology is poorly understood and hence its treatment remains to be established. Intramuscular injections of botulinum toxin type A (BT-A) have also been demonstrated to reduce HSP. The mechanism whereby intramuscular inoculation of BT-A reduces pain may include a muscle relaxant effect and inhibition of the release of neurotransmitters by sensory neurons. Nevertheless, this approach has some limitations: it is probably more effective in muscular than in articular pain and it may be influenced by the muscles affected and site of injection. Intra-articular injection of BT-A has recently proven safe and effective in the treatment of refractory joint shoulder pain caused by chronic arthritis. The mechanisms by which it exerts this effect are not known, but could include inhibition of the release of pain peptides from nerve terminals and sensory ganglia, and anti-inflammatory and anti-glutaminergic effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiparesis and shoulder pain due to first stroke (ischemic or hemorrhagic) admitted in a rehabilitative department to carry out a standard post-acute rehabilitative program
* Pain score of 45 or greater on a 0-100 mm pain visual analog scale (VAS; 0 = no pain, 100 = worst possible pain)
* Duration of HSP for at least one month
* Pain refractoriness to conventional treatment i.e. common analgesics (such as paracetamol and NSAIDs), slings, strapping and handling of the arm, functional electrical stimulation of shoulder muscles

Exclusion Criteria:

* Significant spasticity in the upper shoulder joint, defined as a score of 2 or more at the modified Ashworth scale
* History of shoulder pain or shoulder diseases.
* History of neurological diseases (i.e. Parkinson disease, dystonia).
* History of botulinum toxin treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic superiority of BTA respect steroid in HSP, in patients with hemiparesis and shoulder pain due to stroke (ischemic or hemorrhagic). | one year
  The primary efficacy outcome will be the reduction in pain severity, measured by VAS score after 4 weeks of treatment, with respect to baseline evaluation.
  A difference of about 10 mm between treatments, in the reduction of pain severity, as measured by a VAS scale after 4 weeks, will be considered as clinically significant.

SECONDARY OUTCOMES:
Improvement of upper limb functions and activity | one year
  The secondary efficacy outcome will include the following measures: VAS score at the other time points of the study (1 week, 2 weeks, 3 months and 6 months after the treatment), Shoulder Pain and Disability Index (SPADI), Modified Ashworth Scale (MAS), Fugl Meyer Assessment Scale (FMAS), NIH Stroke Scale index (NISS), Functional Independent Measure (FIM), quality of life on short-form (SF)-36 subscales (SF-36).
Improvement of quality of life | one year
  The secondary efficacy outcome will include the following measures: VAS score at the other time points of the study (1 week, 2 weeks, 3 months and 6 months after the treatment), Shoulder Pain and Disability Index (SPADI), Modified Ashworth Scale (MAS), Fugl Meyer Assessment Scale (FMAS), NIH Stroke Scale index (NISS), Functional Independent Measure (FIM), quality of life on short-form (SF)-36 subscales (SF-36).
Safety Variables | one year
  Safety will be assessed through the collection of adverse events (AEs) and changes in the strength of the deltoid, trapezium, biceps and triceps muscles.
  All treated patients, no matter the duration of treatment, will be considered for the safety analysis.
  Adverse events will be fully described and presented in frequency tables whereas changes in the strength of abovementioned muscles will be summarised by descriptive statistics (mean, standard deviation, minimum and maximum), for the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Galardi, Dr, Study Director — San Raffaele-Giglio Foundation
Locations (1):
- Fondazione Istituto San Raffaele G. Giglio di Cefalù, Cefalù, Palermo, Italy